CLINICAL TRIAL: NCT01373021
Title: Assessment of the Effect of Dexmedetomidine in the Management of Postoperative Pain When Combined With Fentanyl in the Patient-controlled Analgesia
Brief Title: The Effect of Dexmedetomidine on Postoperative Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yong Chul Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: sunrud1129
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Colon Cancer, Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Fentanyl; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- F (Placebo Comparator): Fentanyl+Normal saline
  Interventions: Drug: Fentanyl
- D (Experimental): Fentanyl+Dexmedetomidine
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Fentanyl — Fentanyl 2500mcg+NS50ml
  Arms: F
Drug: Dexmedetomidine — Fentanyl 2500mcg+Dexmedetomidine 500mcg + NS 45ml
  Arms: D

SUMMARY:
The purpose of this study is to determine whether additional Dexmedetomidine to patient controlled analgesia can reduce fentanyl consumption.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery for colon cancer

Exclusion Criteria:

* Liver disease
* Kidney disease
* Allergy for study drugs
* Inability to receive patient controlled analgesia

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
total amount of administered fentanyl | during first 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea